CLINICAL TRIAL: NCT04877353
Title: Postoperative Noninvasive Ventilation After Upper Abdominal Surgery in Chronic Obstructive Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed, PhD candidate _anesthesia ,ICU &pain management_Qena SVU, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIV _COPD
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Acute Respiratory Failure Post Surgical (Diagnosis)
Keywords: noninvasive ventilation; COPD; acute respiratory failure
MeSH Terms: conditions — Disease; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Postoperative NIV
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Experimental): 50 patients.NIV applied for approximately 30 to 45 min at 2- to 4-h intervals for 48 h following surgery
  Interventions: Device: NIV
- group C (No Intervention): 50 patients recieved conventional oxygen therpy.

INTERVENTIONS:
Device: NIV — NIV applied for approximately 30 to 45 min at 2- to 4-h intervals for 48 h following surgery
  Arms: Group N

SUMMARY:
In Qena university hospital a prospective, randomized study was carried out on 100 COPD patients, all were divided into; conventional therapy without NIV (C group) 50 patients or with prophylactic NIV(N group) 50 patients.NIV applied for approximately 30 to 45 min at 2- to 4-h intervals for 48 h following surgery . Primary endpoint was the acute respiratory events (ARE) .Secondary endpoints were acute respiratory failure (ARF), intubation rate, mortality rate, infectious and non-infectious complications, and ICU stay.

ELIGIBILITY:
1. Inclusion criteria:

   * Age˃18 years, scheduled for upper abdominal surgery under general anesthesia.
   * Moderate to very severe COPD (GOLD II to IV).
   * ASA functional status II or greater.
2. Exclusion criteria:

   * Contraindications to the application of NIV.
   * Sleep apnea syndrome.
   * Facial deformation.
   * Inability to follow the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
acute respiratory events | 28days
  patients %

SECONDARY OUTCOMES:
acute respiratory failure | 28 days
  patients %
intubation rate | 28 days
  patients %
ICU mortality | 28 days
  patients %
ICU length of stay | 28 days
  days
infectious and non infectious complications | 28 days
  patients %

CONTACTS AND LOCATIONS:
Locations (1):
- asmaa Mostafa, Luxor, Egypt

IPD SHARING:
Plan to Share IPD: No